CLINICAL TRIAL: NCT00801385
Title: A Multicenter, Open-label, Phase II Study of Sorafenib in Combination With Erlotinib in Non-small Cell Lung Cancer (NSCLC) Refractory to One or Two Prior Chemotherapy Regimens
Brief Title: Sorafenib and Erlotinib in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer That Has Not Responded to Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000618003; YONSEI-4-2008-0160
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Sorafenib; Polymerase Chain Reaction; Immunohistochemistry

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: sorafenib tosylate
Genetic: DNA analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: protein analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Sorafenib and erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Giving sorafenib together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sorafenib together with erlotinib works in treating patients with stage IIIB or stage IV non-small cell lung cancer that has not responded to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response rate of sorafenib tosylate in combination with erlotinib hydrochloride in patients with stage IIIB-IV non-small cell lung cancer refractory to 1 or 2 prior chemotherapy regimens.

Secondary

* To assess the response duration in patients treated with this regimen.
* To assess the disease control rate in patients treated with this regimen.
* To assess the progression-free survival of patients treated with this regimen.
* To assess the overall survival of patients treated with this regimen.
* To assess the safety and tolerability of this regimen in these patients.
* To analyze biomarkers, including evaluation of EGFR expression, mutational analysis of EGFR and K-ras, and immunohistochemical analysis of EGFR downstream pathway (phospho-EGFR, phospho-AKT, phospho-Erk, phospho-STAT3).

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily and oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Tissue samples are analyzed at the nucleic acid level for EGFR mutation (exon 18-21) and K-ras mutation (exon 2), DNA mutations via PCR, presence of EGFR protein by IHC, and downstream effectors of EGFR activation by IHC.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Advanced (stage IIIB-IV) or recurrent disease
* Must have failed 1 or 2 prior chemotherapy regimens, including platinum-containing regimen
* At least 1 unidimensionally measurable lesion > 10 mm by spiral CT scan or > 20 mm by conventional CT scan

  * Previously irradiated lesions cannot be included as sites of measurable disease unless clear tumor progression has been documented in the lesions since the end of radiotherapy
* No known or suspected brain metastases

  * Patients with clinical signs or symptoms that are suspicious of brain metastasis must have a pre-treatment CT scan or MRI of the brain
  * Patients with prior brain metastases are eligible provided they have completed their treatment for brain metastases, no longer require corticosteroids, and are asymptomatic

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC 4,000-12,000/μL
* Neutrophil ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.0 times ULN
* Alkaline phosphatase ≤ 2.0 times ULN
* Serum creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* No active clinically serious infections
* No prior or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1), or any cancer curatively treated > 5 years before study
* Able to swallow oral medications
* No substance abuse or medical, psychological, or social conditions that may interfere with participation in the study or evaluation of the study results

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No prior anti-EGFR targeted therapy
* At least 4 weeks since prior surgery
* At least 4 weeks since prior and no concurrent radiotherapy

  * No prior radiotherapy to the whole pelvis or chest or to ≥ 25% of the bone marrow
* No other concurrent anticancer agents (e.g., chemotherapy or immunotherapy agents) which might affect evaluation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Tumor response based on RECIST criteria

SECONDARY OUTCOMES:
Response duration in patients with confirmed objective response
Disease control rate
Overall survival
Progression-free survival
Biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lim SM, Cho BC, Kim SW, Kang SY, Heo DS, Kim HT, Lee DH, Kim DW, Jung M, Choi JH, Shim HS, Choi JR, Kim JH. A multicenter phase II study of sorafenib in combination with erlotinib in patients with advanced non-small cell lung cancer (KCSG-0806). Lung Cancer. 2016 Mar;93:1-8. doi: 10.1016/j.lungcan.2015.12.005. Epub 2015 Dec 29. PMID 26898607